CLINICAL TRIAL: NCT04145427
Title: Impact of a Low Carbohydrate Diet (LCD) on Metabolic Inflexibility and Cardiovascular Risk in Liver Transplant (LT) Patients
Brief Title: Impact of a LCD on Metabolic Inflexibility and Cardiovascular Risk in Liver Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20017667
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Weight Gain
Keywords: Liver Transplant, Low Carbohydrate Diet
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): This arm will be randomized to low carbohydrate diet
  Interventions: Behavioral: LCD
- Standard Dietary Advice Control Group (Active Comparator): This arm will be randomized to control diet
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Initial Weight Loss consultation
  1.5 hour session on how to do implement healthy diet and then have a 2-week follow-up class. Information on how to maintain a healthy combination protein, fat and vegetables daily will be provided provided.
  4 lifestyle coaching sessions
  Monthly visits for behavioral and dietary coaching as well as medication management.
  Arms: Standard Dietary Advice Control Group
Behavioral: LCD — Initial Weight Loss consultation
  1.5 hour session on how to do implement healthy diet and then have a 2-week follow-up class. Information on how to maintain a LCD will be provided provided.
  4 lifestyle coaching sessions
  Monthly visits for behavioral and dietary coaching as well as medication management.
  Arms: Low Carbohydrate Diet

SUMMARY:
This study is looking to see how a 6-month low carbohydrate diet can affect the body's ability to use energy in addition to the affects it has on the heart and blood vessel health.

DETAILED DESCRIPTION:
Weight gain often occurs following a liver transplant. This weight gain is problematic as it leads to many other health problems. The reasons of this weight gain are still poorly understood. To better understand weight gain, this study is looking to see how a 6-month low carbohydrate diet can affect the body's ability to use energy in addition to the affects it has on heart and blood vessel health.

This study will help researchers to better understand weight gain after a transplant. This knowledge will help doctors prevent weight gain after a liver transplant and therefore improve the health of liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* At least 12 months after LT
* Obese (BMI > 30kg/m2)

Exclusion Criteria:

* Acute cellular or chronic rejection within 3 months
* Post-LT liver or non-liver related malignancy
* Active viral hepatitis (B or C), autoimmune hepatitis
* Untreated biliary strictures or vascular complications (i.e. hepatic artery thrombosis)
* Poorly controlled Diabetes mellitus
* Relapse of alcohol abuse after LT
* Stage 5 Chronic Kidney Disease
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in weight | baseline to 6 months
  Weight will be measured on a standardized scale in kilograms that will be zeroed out prior to the measurement

SECONDARY OUTCOMES:
Change in metabolic flexibility | baseline to 6 months
  This will be measured in whole room calorimeter and reported as respiratory quotient
Change in LDL-C | baseline to 6 months
  LDL-cholesterol will be measured using a fasting blood draw and a standard lipid panel.
Change in total cholesterol | baseline to 6 months
  Total cholesterol will be measured using a fasting blood draw and a standard lipid panel.
Change in small dense low-density lipoprotein | baseline to 6 months
  Small dense LDL will be measured using a fasting blood draw and a standard lipid panel.
Change in adiposity | baseline to 6 months
  This will be measured on body composition MRI where subcutaneous and visceral fat will be quantified. Subcutaneous fat and visceral fat volume will measured on body composition MRI in liters (L) and standardized to body height and will be reported as liter/m2

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Siddiqui, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No